CLINICAL TRIAL: NCT00005036
Title: A Randomized Phase III Equivalence Trial of Irinotecan (CPT-11) Versus Oxaliplatin (OXAL)/5-Fluorouracil (5-FU)/Leucovorin (CF) in Patients With Advanced Colorectal Carcinoma Previously Treated With 5-FU
Brief Title: Irinotecan Compared With Combination Chemotherapy in Treating Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: SWOG Cancer Research Network (Network); Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01847; N9841; SWOG-N9841; NCCTG-N9841; CDR0000067623; ECOG-N9841; U10CA025224 (NIH)
Record Dates: First submitted 2000-04-06; First posted 2003-01-27 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Mucinous Adenocarcinoma of the Colon; Mucinous Adenocarcinoma of the Rectum; Recurrent Colon Cancer; Recurrent Rectal Cancer; Signet Ring Adenocarcinoma of the Colon; Signet Ring Adenocarcinoma of the Rectum; Stage IIIA Colon Cancer; Stage IIIA Rectal Cancer; Stage IIIB Colon Cancer; Stage IIIB Rectal Cancer; Stage IIIC Colon Cancer; Stage IIIC Rectal Cancer; Stage IVA Colon Cancer; Stage IVA Rectal Cancer; Stage IVB Colon Cancer; Stage IVB Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Irinotecan; Oxaliplatin; Leucovorin; Fluorouracil

ARMS (2):
- Arm I (irinotecan) (Experimental): Patients receive irinotecan IV over 90 minutes on day 1. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: irinotecan hydrochloride; Procedure: quality-of-life assessment
- Arm II (oxalipatin, fluorouracil, leucovorin calcium) (Experimental): Patients receive oxaliplatin IV over 2 hours on day 1, leucovorin calcium IV over 2 hours on days 1 and 2, and fluorouracil IV bolus followed by IV infusion over 22 hours on days 1 and 2. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: oxaliplatin; Drug: leucovorin calcium; Drug: fluorouracil; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E
  Arms: Arm I (irinotecan)
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
  Arms: Arm II (oxalipatin, fluorouracil, leucovorin calcium)
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
  Arms: Arm II (oxalipatin, fluorouracil, leucovorin calcium)
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
  Arms: Arm II (oxalipatin, fluorouracil, leucovorin calcium)
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
Randomized phase III trial to compare the effectiveness of irinotecan with that of combination chemotherapy in treating patients who have advanced colorectal cancer that has not responded to previous treatment. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which chemotherapy regimen is more effective for colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine whether in advanced colorectal carcinoma patients who have been previously treated with 5-FU, the overall survival of patients treated with OXAL + 5-FU + CF followed by CPT-11 is equivalent to the survival of patients treated with CPT-11 followed by OXAL + 5-FU + CF.

SECONDARY OBJECTIVES:

I. Evaluation of time to tumor progression, time to treatment failure, toxicity of treatment, and overall response rate in patients treated with these two regimens.

II. To compare quality-of-life measurements patients treated with these two regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to performance status (ECOG 0-1 vs 2), primary indicator lesion (hepatic vs pulmonary vs other), age (less than 65 vs at least 65 years), alkaline phosphatase (less than 2 vs at least 2 times ULN), fluorouracil failure (adjuvant vs metastatic), and membership (intergroup vs expanded participation project). Patients are randomized to one of two treatment arms.

ARM I: Patients receive irinotecan IV over 90 minutes on day 1. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive oxaliplatin IV over 2 hours on day 1, leucovorin calcium IV over 2 hours on days 1 and 2, and fluorouracil IV bolus followed by IV infusion over 22 hours on days 1 and 2. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity.

Patients who experience progression or toxicity on the initial regimen may crossover to the other regimen. At least 3 weeks must elapse between regimens.

Quality of life is assessed at baseline, prior to each chemotherapy course, at crossover, and at the end of the study.

Patients are followed every 6 months for 3 years or until death.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced, locally recurrent,or metastatic colorectal adenocarcinoma not curable by surgery or radiotherapy
* Progressive disease following:

  * One prior fluorouracil based chemotherapy regimen for metastatic disease
  * Failure during or within 6 months after fluorouracil based adjuvant therapy
* Measurable or evaluable disease
* No CNS metastases or carcinomatous meningitis
* Performance status - ECOG 0-2
* At least 12 weeks
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL (transfusion allowed)
* Bilirubin no greater than 1.5 mg/dL
* AST no greater than 5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 5 times ULN
* Creatinine no greater than 1.5 times ULN
* No uncontrolled high blood pressure
* No unstable angina
* No symptomatic congestive heart failure
* No myocardial infarction with the past 6 months
* No serious uncontrolled cardiac arrhythmias
* No New York Heart Association class III or IV heart disease
* No pleural effusion or ascites that cause respiratory compromise (e.g., dyspnea grade 2 or greater)
* No interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Fluent in English
* No active or uncontrolled infection
* No other prior malignancy within the past 5 years, except:
* Adequately treated basal or squamous cell skin cancer
* Adequately treated noninvasive carcinomas
* No sensory neuropathy grade 2 or greater
* No uncontrolled colonic or small bowel disorders (greater than 3 loose stools daily)
* No concurrent sargramostim (GM-CSF)
* At least 4 weeks since prior chemotherapy and recovered
* No more than 1 prior chemotherapy regimen for advanced colorectal cancer
* No prior irinotecan or other camptothecin derivative (e.g., topotecan)
* No prior oxaliplatin
* No other concurrent investigational chemotherapy agents
* At least 4 weeks since prior major radiotherapy
* No prior radiotherapy to greater than 25% of bone marrow
* At least 4 weeks since prior major surgery and recovered
* At least 2 weeks since prior minor surgery and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 1999-11; Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | At least 6 months
  The primary analysis for this trial will be based on a one-sided Generalized Wilcoxon test.

SECONDARY OUTCOMES:
Time-to-tumor progression | Time from start of therapy to documentation of disease progression, assessed up to 3 years
Time-to-treatment failure | Time from the date of randomization to the date at which the patient is removed from treatment due to progression, toxicity, refusal, or death, assessed up to 3 years
Objective tumor response rate (CR or PR) in patients with measureable disease | At least 4 weeks
Toxicity and dose intensity | Up to 3 years
Quality of life | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Henry Pitot, Principal Investigator — North Central Cancer Treatment Group
Locations (1):
- North Central Cancer Treatment Group, Rochester, Minnesota, United States